CLINICAL TRIAL: NCT02592707
Title: An International, Multicenter, Open-label Study to Evaluate Safety, Tolerability, Biodistribution, Dosimetry and Preliminary Efficacy of 177Lu-OPS201 for the Therapy of Somatostatin Receptor-positive Neuroendocrine Tumors (NETs)
Brief Title: Study to Evaluate the Safety and Preliminary Efficacy of 177Lu-OPS201 in NETs
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated (Due to small number of ongoing patients. Patients ongoing at time of termination could choose to join study D-FR-01072-004 for long term follow-up.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D-FR-01072-001; 2015-002867-41 (EudraCT Number); OPS-C-001 (Other: Initial sponsor study ID)
Record Dates: First submitted 2015-10-15; First posted 2015-10-30 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 177Lu-DOTA-JR11; amino-acid, glucose, and electrolyte solution; arginyllysine; Antiemetics; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 177Lu-IPN01072 (Experimental): 177Lu-IPN01072 administered in 3 cycles at intervals of 8 weeks (+ up to 2 additional optional cycles)
  Interventions: Drug: Satoreotide tetraxetan; Other: Amino acid solution; Other: Antiemetic

INTERVENTIONS:
Drug: Satoreotide tetraxetan — Satoreotide tetraxetan administered in 3 cycles at intervals of 8 weeks (+ up to 2 additional optional cycles)
  Other Names: 177Lu-OPS201; 177Lu-IPN01072
Other: Amino acid solution — Given as an auxiliary product the day of the IMP infusion for safety reasons to protect the renal function.
  Centres can use their established amino acid infusion or Ipsen amino acid solution (auxiliary medical product OPS301)
  Other Names: OPS301; IPN60070; Arginine and lysine
Other: Antiemetic — To counteract the known side effects of the amino acid infusion, such as nausea, dexamethasone (antiemetic) and as-required ondansetron will be administered 15 to 30 minutes before the start of the amino acid infusion (unless there are contraindications for these drugs).
  Other Names: Dexamethasone; Ondansetron

SUMMARY:
The purpose of this clinical phase I/II study was to investigate the safety and tolerability of satoreotide tetraxetan (177Lu-IPN01072, formerly known as 177Lu-OPS201) used for the treatment of patients with neuroendocrine tumors (NETs). The secondary objectives of this study were the assessment of biodistribution, dosimetry and preliminary efficacy of satoreotide tetraxetan.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Patients of either gender, aged ≥ 18 years.
3. Women of childbearing potential (not surgically sterile or less than 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 6 months after the last dose. Acceptable methods of contraception include abstinence, or double contraception: steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method (intrauterine device, condom etc.).
4. Male patients must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 6 months after the last activity administration.
5. Karnofsky performance score ≥ 60.
6. Life expectancy of at least 6 months.
7. Histologically confirmed diagnosis of -

   * unresectable GEP NET (Grade I and Grade II according to WHO classification (2010, Annex 01), functioning and non-functioning).
   * unresectable "typical lung carcinoid" or "atypical lung carcinoid" are acceptable (with the exception of Large Cell Bronchial Neuroendocrine Neoplasms and Small Cell Lung Cancers) (Caplin 2015).
   * malignant, unresectable pheochromocytoma or paraganglioma
8. Documentation of progressive disease based on RECIST v1.1 under prior anti-tumor therapy within 6 months of entry in the study (although the progression might have occurred more than 6 months before study entry). Patients should not have received further anti-tumor therapy once disease progression is documented. The images of this evaluation should be available for TGR evaluation.
9. In countries where sunitinib or everolimus are marketed, patients with GEP NET and lung NET will be progressive under this prior anti-tumor treatment for the respective indication. Patients not suitable for everolimus/sunitinib therapy according to a tumor board decision (or comparable local practice) may also be enrolled into the study. Patients having everolimus/sunitinib therapy should have a wash-out phase of ≥ 4 weeks before the first treatment.
10. Measurable disease based on RECIST v1.1.
11. Confirmed presence of somatostatin receptors on technically evaluable tumor lesions documented by a positive Somatostatin Receptor Scan performed within 6 months prior to enrolment in the study.
12. Calculated GFR ≥ 55 mL/min.
13. Blood test results as follows:

    * Leukocytes: ≥ 4*10^9/L
    * Erythrocytes: ≥ 3.5*12^9/L
    * Platelets: ≥ 100*10^9/L
    * Albumin: > 30 g/L
    * ALT, AST, AP: ≤ 5 times ULN (upper limit of normal)
    * Bilirubin: ≤ 2 times ULN (2x 1.1 mg/dL)

Exclusion Criteria:

1. Known hypersensitivity to 177Lu, to DOTA, to JR11 or to any of the excipients of 177Lu-OPS201.
2. Any previous peptide receptor radionuclide therapy (PRRT).
3. Diagnosis of thymic NET.
4. Presence of active infection at screening or history of serious infection within the previous 6 weeks.
5. Administration of any other investigational medicinal product within 60 days prior to entry.
6. Prior or planned administration of a therapeutic radiopharmaceutical within 8 half-lives of the radionuclide including any time during the current study.
7. Any extensive radiotherapy ≤ 3 months before enrolment.
8. Chemotherapy ≤ 3 months before enrolment.
9. Nephrectomy, renal transplant or concomitant nephrotoxic therapy putting the subject at high risk of renal toxicity during the study as assessed by the investigator.
10. Pregnant or breast-feeding women: A pregnancy test will be performed at the start of the study for all female patients of childbearing potential (i.e. not surgically sterile or up to 2 years postmenopausal).
11. Any uncontrolled significant medical, psychiatric or surgical condition (active infection, unstable angina pectoris, cardiac arrhythmia, poorly controlled hypertension, poorly controlled diabetes mellitus [HbA1c ≥9%], uncontrolled congestive heart disease, etc.) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety or that would limit compliance with the objectives and assessments of the study. Note: the patient should be able to tolerate high volume load.
12. Current history of any malignancy other than NET within 5 years of enrolment except for fully -resected non-melanoma skin cancer or cervical cancer in situ. Current history of malignancy; patients with a secondary tumor in remission of > 5 years can be included
13. Any mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- MD Anderson Cancer Center, Department of Nuclear Medicine, Houston, Texas, United States
- Australia (2):
  - Peter MacCallum Cancer Centre, Molecular Imaging and Targeted Therapeutics Laboratory, East Melbourne
  - Ramsay Hollywood Private Hospital, Department of Nuclear Medicine, Perth
- University Hospital Vienna, Department of Nuclear Medicine, Vienna, Austria
- CHU de Quebec - Universite Laval Research Center, Department of Radiology and Nuclear Medicine, Québec, Canada
- University Hospital Aarhus, Department of Hepatology and Gastroenterology, Aarhus, Denmark
- CHU de Nantes, Hotel Dieu, Service de Medecine Nucleaire, Nantes, France
- University Hospital Basel, Department of Nuclear Medicine, Basel, Switzerland
- Royal Free Hospital, Department of Nuclear Medicine, London, United Kingdom

REFERENCES:
- [Derived] Schurrle SB, Eberlein U, Ansquer C, Beauregard JM, Durand-Gasselin L, Gronbaek H, Haug A, Hicks RJ, Lenzo NP, Navalkissoor S, Nicolas GP, Pais B, Volteau M, Wild D, McEwan A, Lassmann M. Dosimetry and pharmacokinetics of [177Lu]Lu-satoreotide tetraxetan in patients with progressive neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2024 Jul;51(8):2428-2441. doi: 10.1007/s00259-024-06682-1. Epub 2024 Mar 26. PMID 38528164
- [Derived] Wild D, Gronbaek H, Navalkissoor S, Haug A, Nicolas GP, Pais B, Ansquer C, Beauregard JM, McEwan A, Lassmann M, Pennestri D, Volteau M, Lenzo NP, Hicks RJ. A phase I/II study of the safety and efficacy of [177Lu]Lu-satoreotide tetraxetan in advanced somatostatin receptor-positive neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2023 Dec;51(1):183-195. doi: 10.1007/s00259-023-06383-1. Epub 2023 Sep 18. PMID 37721581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/2, open-label study was conducted in participants with somatostatin receptor positive neuroendocrine tumour (NETs) at 8 investigational sites in Australia, Austria, Canada, Denmark, France, Switzerland and United Kingdom between 06 March 2017 and 22 February 2022. The sponsor terminated the study early for strategic reasons and this decision was not due to any safety or tolerability concern of the study drug.
Pre-assignment Details: The study was performed in 2 parts, Part A and Part B. Study consists of a screening period (up to 4 weeks), Treatment period (3 core treatment cycles in each Part A and Part B; 2 additional cycles in Part B only) and followed by long-term follow-up (LTFU) period (2 years). Each cycle was 8 weeks (+ up to 4 weeks if toxicity) apart. A total 40 participants were treated in this study. Due to initial findings, Cohorts 2, 4, 5, 7 and 8 in Part B were not performed in this study.
Groups:
- Part A: 177Lu-IPN01072 4.5 GBq: Participants received 4.5 gigabecquerel (GBq) 177Lu-IPN01072 [target dose of 300 microgram (mcg) ±50 mcg] intravenous (IV) infusion on Day 1 of 3 treatment cycles. Each cycle was 8 weeks apart [+2 weeks or up to +4 weeks in case of adverse events (AE) which had not adequately recovered].
- Part B Cohort 1: 177Lu-IPN01072 6 GBq: Participants received 6 GBq 177Lu-IPN01072 (target dose of 300 mcg) IV infusion on Day 1 of 3 treatment cycles. The radioactivity dose was reduced to 4.5 GBq in Cohort 1 adapted as recommended by data review board (DRB). As a result, Cohort 1 adapted was similar to Cohort 1 except the radioactivity dose was 4.5 GBq. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Part B Cohort 3: 177Lu-IPN01072 4.5 GBq: Participants received 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg in Cycle 1; 700 mcg in Cycle 2; 300 mcg in Cycle 3) IV infusion on Day 1 of 3 treatment cycles. Target dose was 300 mcg for additional cycles, if any. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Part B Cohort 6: 177Lu-IPN01072 4.5 GBq: Participants received of 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg in Cycle 1; 1300 mcg in Cycle 2; 300 mcg in Cycle 3) IV infusion on Day 1 of 3 treatment cycles. Target dose was 300 mcg for additional cycles, if any. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
Period: Overall Study
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq
Started | 15 | 6 | 9 | 10
Completed (Completed LTFU period) | 9 | 1 | 3 | 3
Not Completed | 6 | 5 | 6 | 7
Not completed — Consent Withdrawn | 0 | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 4 | 4 | 3 | 3
Not completed — Other | 0 | 0 | 1 | 2
Not completed — Never entered LTFU period | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all participants who received 177Lu-IPN01072.
Groups:
- Part A: 177Lu-IPN01072 4.5 GBq: Participants received 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg ±50 mcg) IV infusion on Day 1 of 3 treatment cycles. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AE which had not adequately recovered).
- Part B Cohort 1: 177Lu-IPN01072 6 GBq: Participants received 6 GBq 177Lu-IPN01072 (target dose of 300 mcg) IV infusion on Day 1 of 3 treatment cycles. The radioactivity dose was reduced to 4.5 GBq in Cohort 1 adapted as recommended by DRB. As a result, Cohort 1 adapted was similar to Cohort 1 except the radioactivity dose was 4.5 GBq. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Total: Total of all reporting groups
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | Total
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (12.9) | 65.3 (8.9) | 55.0 (16.0) | 56.7 (13.7) | 59.9 (13.5)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 7 | 3 | 6 | 7 | 23
  >=65 | 8 | 3 | 3 | 3 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 3 | 6 | 19
  Male | 7 | 4 | 6 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 6 | 9 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 15 | 6 | 9 | 9 | 39
  Other | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: AE is defined as any untoward medical occurrence in a subject or clinical trial subject administered a medicinal product, which did not necessarily have a causal relationship with this treatment. A serious AE (SAE) was classified as any untoward medical occurrence that at any dose results in death; AE was life threatening; required inpatient hospitalization or prolonged existing hospitalization; resulted in persistent or significant disability/ incapacity; was a congenital anomaly/birth defect; was an important medical event that may not result in death. TEAEs are defined as AEs that developed or worsened after start of treatment.
Time Frame: From the start of the first study medication (Cycle 1 Day 1) up to 6 months after the last dose of study medication, maximum of 33 months
Population: The SAS included all participants who received 177Lu-IPN01072.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Participants who received 177Lu-IPN01072 dose from 4.5 to 6 GBq (target dose of 300 to 1300 mcg) as IV infusion on Day 1 of 3 treatment cycles/additional 2 cycles (when applicable). Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AE which had not adequately recovered).
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
Participants
  TEAEs | 15 | 6 | 9 | 10 | 40
  Serious TEAEs | 2 | 1 | 2 | 3 | 8

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: DLTs were defined as study medication-related AEs with a severity of Grade 3 or higher are considered DLT, with the exception of hair loss, lymphopenia, nonfebrile neutropenia lasting <4 weeks and thrombocytopenia lasting <4 weeks.
Time Frame: From the start of the first study medication (Cycle 1 Day 1) up to EOCT, maximum of 16 weeks.
Population: The SAS included all participants who received 177Lu-IPN01072.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
Participants | 3 | 0 | 2 | 1 | 6

3. Secondary Outcome: Maximum Uptake (%) of 177Lu-IPN01072 at Target Lesions and Discernible Organs in Cycle 1
Description: 177Lu-IPN01072 uptake in organs and lesions was evaluated centrally, using nuclear medicine images, as part of the dosimetry workflow. Uptake activity for organs of interest (i.e., body, bone marrow, kidney [left + right], healthy liver, and spleen) was determined. The maximal uptake in lesions was calculated for each lesion as: maximal activity divided injected activity*100.
Time Frame: 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: The Per Protocol Dosimetry Analysis Set (PP-DAS) included all participants in the Intent-To-Treat Dosimetry Analysis Set (ITT-DAS) for whom no major protocol violations occurred affecting dosimetry variables. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: percentage of injected drug activity
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 11 | 6 | 9 | 10 | 36
percentage of injected drug activity
  Bone marrow (image-based): number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
  Bone marrow (image-based) | 0.0469 [0.0246 to 0.0751] | 0.0420 [0.0100 to 0.280] | 0.0250 [0.0149 to 0.0570] | 0.0219 [0.0053 to 0.0300] | 0.0380 [0.0053 to 0.280]
  Liver: number analyzed (Participants) | 7 | 1 | 0 | 0 | 8
  Liver | 1.52 [0.314 to 6.34] | 4.31 [4.31 to 4.31] |  |  | 2.63 [0.314 to 6.34]
  Kidney (left + right): number analyzed (Participants) | 11 | 6 | 9 | 9 | 35
  Kidney (left + right) | 1.96 [0.980 to 3.82] | 1.76 [1.05 to 2.08] | 1.60 [1.19 to 2.51] | 1.67 [0.749 to 2.41] | 1.76 [0.749 to 3.82]
  Spleen: number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
  Spleen | 1.50 [0.274 to 2.93] | 1.27 [0.960 to 2.46] | 1.78 [0.550 to 5.97] | 1.79 [1.19 to 2.65] | 1.67 [0.274 to 5.97]
  All lesions: number analyzed (Participants) | 11 | 5 | 9 | 8 | 33
  All lesions | 0.651 [0.0290 to 6.35] | 2.36 [0.266 to 8.74] | 1.18 [0.235 to 18.7] | 1.43 [0.190 to 15.0] | 0.932 [0.0290 to 18.7]

4. Secondary Outcome: Maximal Uptake (%) of 177Lu-IPN01072 in Blood in Cycle 1
Description: 177Lu-IPN01072 uptake in blood was evaluated on site/locally using a gamma counter calibrated for 177Lu-IPN01072 according to the dosimetry operational manual.
Time Frame: Pre-infusion (Baseline), 5 and 30 minutes, 1, 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: The radiopharmaceutical pharmacokinetic (PK) set included all participants in the ITT set who received at least 1 dose of study medication and had at least 1 measured radioactive concentration in blood. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: percentage/liter (L)
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 6 | 8 | 10 | 37
percentage/liter (L) | 3.66 [2.17 to 7.88] | 2.98 [2.26 to 4.35] | 2.77 [1.98 to 7.35] | 3.32 [0.539 to 4.11] | 3.03 [0.539 to 7.88]

5. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of 177Lu-IPN01072 in Discernible Organs in Cycle 1
Description: The AUC of 177Lu-IPN01072 radioactivity in discernible organs were computed for each administration of 177Lu-IPN01072.
Time Frame: 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: The PP-DAS included all participants in the ITT-DAS for whom no major protocol violations occurred affecting dosimetry variables. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: MBq*hour
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 11 | 6 | 9 | 10 | 36
MBq*hour
  Bone marrow (Image-based): number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
  Bone marrow (Image-based) | 174 [45.3 to 224] | 352 [154 to 3988] | 138 [91.0 to 362] | 157 [41.5 to 244] | 175 [41.5 to 3988]
  Kidney (left + right): number analyzed (Participants) | 11 | 6 | 9 | 9 | 35
  Kidney (left + right) | 9596 [3896 to 26596] | 8966 [7350 to 10586] | 6239 [5853 to 11269] | 7578 [3320 to 9815] | 8239 [3320 to 26596]
  Liver: number analyzed (Participants) | 7 | 1 | 0 | 0 | 8
  Liver | 6745 [755 to 20751] | 17918 [17918 to 17918] |  |  | 11133 [755 to 20751]
  Spleen: number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
  Spleen | 6701 [1134 to 21451] | 7949 [4945 to 11734] | 7727 [1547 to 28269] | 8179 [3901 to 12355] | 7772 [1134 to 28269]

6. Secondary Outcome: AUC of 177Lu-IPN01072 in Blood in Cycle 1
Description: The AUC of 177Lu-IPN01072 radioactivity in blood were computed for each administration of 177Lu-IPN01072.
Time Frame: Pre-infusion (Baseline), 5 and 30 minutes, 1, 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: The radiopharmaceutical PK set included all participants in the ITT set who received at least 1 dose of study medication and had at least 1 measured radioactive concentration in blood. Only data from the participants analyzed were reported.
Measure: Median (Full Range); unit: MBq*hour/L
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 6 | 8 | 10 | 37
MBq*hour/L | 623 [299 to 1003] | 901 [442 to 1806] | 690 [371 to 1201] | 720 [290 to 1034] | 726 [290 to 1806]

7. Secondary Outcome: Terminal Half-Life (T1/2) of Radioactivity Concentrations of the Radiopharmaceutical in Blood in Cycle 1
Description: The terminal half-life was defined as the largest half-life of the decay curve of blood activity.
Time Frame: Pre-infusion (Baseline), 5 and 30 minutes, 1, 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 6 | 8 | 10 | 37
hours | 68.3 [42.2 to 160] | 109 [38.6 to 160] | 123 [41.2 to 160] | 145 [55.3 to 160] | 127 [38.6 to 160]

8. Secondary Outcome: Highest Absorbed Dose of 177LU-IPN01072 to Each Discernible Organ in Cycle 1
Description: The absorbed dose to the discernible organs (i.e., organs showing uptake) was evaluated centrally, using nuclear medicine images, as part of the dosimetry workflow. The organs considered for 177LU-IPN01072 image-based dosimetry assessment included: liver, bone marrow, kidney (left + right), and spleen. Highest absorbed dose of 177Lu-IPN01072 was calculated as described in the Dosimetry calculation procedure manual. Maximum value observed for each discernible organs across participants has been reported.
Time Frame: 4, 24, 48, 72 to 96 and 144 to 168 hours post infusion in Cycle 1
Population: as for outcome 5
Measure: Number; unit: Gray
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 11 | 6 | 9 | 10 | 36
Gray
  Bone marrow (image-based assay): number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
  Bone marrow (image-based assay) | 0.97 | 3.59 | 0.50 | 0.69 | 3.59
  Kidney (left + right): number analyzed (Participants) | 11 | 6 | 9 | 9 | 35
  Kidney (left + right) | 8.55 | 4.87 | 5.86 | 5.07 | 8.55
  Liver: number analyzed (Participants) | 7 | 1 | 0 | 0 | 8
  Liver | 1.26 | 0.81 |  |  | 1.26
  Spleen: number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
  Spleen | 8.07 | 6.00 | 5.90 | 4.09 | 8.07

9. Secondary Outcome: Specific Absorbed Dose Per Organ and Lesions of 177Lu-IPN01072 in Cycle 1
Description: The specific absorbed dose was evaluated centrally, using nuclear medicine images, as part of the dosimetry workflow. Data are presented for all lesions, regardless of their anatomical localization. The organs considered for 177Lu-IPN01072 image-based dosimetry assessment included: liver, bone marrow, kidney (left + right), and spleen. The specific absorbed dose to the lesions was the absorbed dose by the lesion (unit: Gray) divided by the injected radioactivity (unit: GBq) for each lesion selected for dosimetry evaluation. The specific absorbed dose for a given organ was the absorbed dose by this organ (unit: Gray) divided by the injected radioactivity (unit: GBq).
Time Frame: 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycle 1
Population: as for outcome 5
Measure: Median (Full Range); unit: Gray/GBq
Groups:
- Part A: 177Lu-IPN01072 4.5 GBq: Participants received 3 cycles of 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg) on Day 1 of each cycle. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Part B Cohort 1: 177Lu-IPN01072 6 GBq: Participants received 3 cycles of 6 GBq 177Lu-IPN01072 (target dose of 300 mcg) on Day 1 of each cycle. In Cohort 1, there was an adapted radioactivity level and not adapted. In Cohort 1 adapted radioactivity dose was reduced to 4.5 GBq. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Part B Cohort 3: 177Lu-IPN01072 4.5 GBq: Participants received 3 cycles of 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg in Cycle 1; 700 mcg in Cycle 2; 300 mcg in Cycle 3; 300 mcg for additional cycles of 4 and 5) on Day 1 of each cycle. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
- Part B Cohort 6: 177Lu-IPN01072 4.5 GBq: Participants received 3 cycles of 4.5 GBq 177Lu-IPN01072 (target dose of 300 mcg in Cycle 1; 1300 mcg in Cycle 2; 300 mcg in Cycle 3; 300 mcg for additional cycles of 4 and 5) on Day 1 of each cycle. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 11 | 6 | 9 | 10 | 36
Gray/GBq
  Lesions: number analyzed (Participants) | 11 | 5 | 9 | 8 | 33
  Lesions | 2.56 [0.431 to 14.3] | 3.90 [1.92 to 83.3] | 6.82 [2.07 to 28.2] | 13.5 [2.20 to 81.0] | 5.00 [0.431 to 83.3]
  Bone marrow (image-based): number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
  Bone marrow (image-based) | 0.0796 [0.0431 to 0.216] | 0.135 [0.0900 to 0.610] | 0.0850 [0.0700 to 0.110] | 0.0650 [0.0100 to 0.150] | 0.0900 [0.0100 to 0.610]
  Kidney (left + right): number analyzed (Participants) | 11 | 6 | 9 | 9 | 36
  Kidney (left + right) | 1.05 [0.522 to 1.85] | 0.720 [0.600 to 1.02] | 0.880 [0.460 to 1.18] | 0.765 [0.420 to 1.10] | 0.879 [0.420 to 1.85]
  Liver: number analyzed (Participants) | 7 | 1 | 0 | 0 | 8
  Liver | 0.186 [0.146 to 0.279] | 0.170 [0.170 to 0.170] |  |  | 0.179 [0.146 to 0.279]
  Spleen: number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
  Spleen | 0.769 [0.208 to 1.79] | 0.945 [0.500 to 1.08] | 0.985 [0.180 to 1.46] | 0.805 [0.360 to 0.980] | 0.840 [0.180 to 1.79]

10. Secondary Outcome: Cumulative Absorbed Organ Doses of 177Lu-IPN01072 in Cycles 1 and 3
Description: The cumulative absorbed dose to the discernible organs (i.e., organs showing uptake) was evaluated centrally, using nuclear medicine images, as part of the dosimetry workflow.
Time Frame: 4, 24, 48, 72 to 96 hours, 144 to 168 hours post infusion in Cycles 1 and 3
Population: as for outcome 5
Measure: Median (Full Range); unit: Gray
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 11 | 6 | 9 | 10 | 36
Gray
  Cycle 1: Bone marrow (image-based): number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
  Cycle 1: Bone marrow (image-based) | 0.319 [0.102 to 0.974] | 0.715 [0.390 to 3.59] | 0.375 [0.260 to 0.500] | 0.285 [0.0400 to 0.690] | 0.400 [0.0400 to 3.59]
  Cycle 1: Kidney (left + right): number analyzed (Participants) | 11 | 6 | 9 | 9 | 35
  Cycle 1: Kidney (left + right) | 4.31 [2.17 to 8.07] | 3.85 [3.36 to 4.58] | 3.25 [1.79 to 5.34] | 3.55 [1.74 to 4.88] | 3.73 [1.74 to 8.07]
  Cycle 1: Liver: number analyzed (Participants) | 7 | 1 | 0 | 0 | 8
  Cycle 1: Liver | 0.720 [0.336 to 1.26] | 0.810 [0.810 to 0.810] |  |  | 0.765 [0.336 to 1.26]
  Cycle 1: Spleen: number analyzed (Participants) | 9 | 6 | 6 | 6 | 27
  Cycle 1: Spleen | 2.88 [0.844 to 8.07] | 4.35 [3.17 to 6.00] | 4.00 [0.710 to 5.90] | 3.55 [1.48 to 4.09] | 3.45 [0.710 to 8.07]
  Cycle 3: Bone marrow (image-based): number analyzed (Participants) | 11 | 1 | 6 | 3 | 21
  Cycle 3: Bone marrow (image-based) | 1.11 [0.636 to 2.17] | 1.48 [1.48 to 1.48] | 1.09 [0.830 to 1.24] | 0.840 [0.290 to 1.23] | 1.10 [0.290 to 2.17]
  Cycle 3: Kidney (left + right): number analyzed (Participants) | 11 | 1 | 8 | 5 | 25
  Cycle 3: Kidney (left + right) | 12.3 [7.67 to 24.1] | 9.41 [9.41 to 9.41] | 8.91 [6.29 to 14.0] | 10.1 [6.95 to 11.5] | 10.8 [6.29 to 24.1]
  Cycle 3: Liver: number analyzed (Participants) | 7 | 0 | 0 | 0 | 7
  Cycle 3: Liver | 2.08 [1.01 to 4.14] |  |  |  | 2.08 [1.01 to 4.14]
  Cycle 3: Spleen: number analyzed (Participants) | 9 | 1 | 5 | 3 | 18
  Cycle 3: Spleen | 6.93 [4.99 to 15.6] | 7.58 [7.58 to 7.58] | 9.21 [2.82 to 14.6] | 8.08 [5.66 to 14.2] | 8.32 [2.82 to 15.6]

11. Secondary Outcome: Cumulative Amount of Lu-177 Radioactivity Excreted Into the Urine (0 to 48 Hours) [Ae (0-48h)] in Cycle 1
Description: Urine was collected during the first 48 hours post infusion to determine the renal excretion of 177Lu-IPN01072 at Cycle 1 only.
Time Frame: 0 to 6 hours, 6 to 24 hours, 24 to 48 hours post-infusion in Cycle 1 of Part A; 0 to 4 hours, 4 to 24 hours, 24 to 48 hours in Cycle 1 of Part B.
Population: The Radiopharmaceutical PK Set (Part A and Part B) included all participants in the ITT set who received at least 1 dose of study medication and had at least 1 measured radioactive concentration in blood.
Measure: Median (Full Range); unit: Mbq
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 6 | 8 | 9 | 36
Mbq | 2586 [1722 to 4450] | 3106 [2558 to 3998] | 2640 [1346 to 3375] | 2621 [471 to 3181] | 2787 [471 to 4450]

12. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of IPN01072 in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: Pre-infusion (Baseline) and 5 minutes, 30 minutes, 60 minutes, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours after the end of the infusion in Cycle 1
Population: The IPN01072 PK set in plasma (Part B only) included all participants in the ITT set who received at least 1 dose of study medication and have no major protocol deviations affecting the plasma PK variables and who had a sufficient number of plasma levels to estimate the main PK parameters. Only data from the participants analyzed were reported. Results were combined for IPN01072 PK analysis performed at cycle 1, as pre-specified according to study protocol and the data analysis plan.
Measure: Median (Full Range); unit: hours
Groups:
- Part B: All Participants: IPN01072 PK monitoring was performed on cycle 1 only. Participants received 177Lu-IPN01072 dose from 4.5 to 6 GBq (target IPN01072 dose 300 mcg) as IV infusion on Day 1 cycle. The radioactivity dose was reduced to 4.5 GBq in Cohort 1 adapted as recommended by DRB. As a result, Cohort 1 adapted was similar to Cohort 1 except the radioactivity dose was 4.5 GBq. Each cycle was 8 weeks apart (+2 weeks or up to +4 weeks in case of AEs which had not adequately recovered).
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 16
hours | 0.083 [0.00 to 0.28]

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of IPN01072 in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram (ng)/milliliter (mL)
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 16
nanogram (ng)/milliliter (mL) | 10.7 (5.47)

14. Secondary Outcome: AUC From Time Zero to Infinity (AUCinf) of IPN01072 in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*hour (h)/mL
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 15
ng*hour (h)/mL | 45.8 (20.6)

15. Secondary Outcome: T1/2 of IPN01072 in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 15
hours | 6.09 (1.59)

16. Secondary Outcome: Apparent Total Plasma Clearance of IPN01072 (Total CL) in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 15
L/h | 9.58 (12.8)

17. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz) of IPN01072 in Cycle 1
Description: The PK sampling was performed from Day 1 to Day 3 post infusion done at Cycle 1 for Part B only.
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 15
Liter | 68.7 (52.0)

18. Secondary Outcome: Ae (0-48h) of IPN01072 in Cycle 1
Description: Urine was collected during the first 48 hours post infusion to determine the renal excretion of 177Lu-IPN01072 at Cycle 1 for Part B only.
Time Frame: 0 to 4 hours, 4 to 24 hours, 24 to 48 hours in Cycle 1 of Part B
Population: The IPN01072 PK set in urine (Part B only) included all participants in the ITT set who received at least 1 dose of study medication and have no major protocol deviations affecting the urine PK variables and who had all urine IPN01072 levels to estimate the main urine PK parameters. Results were combined for IPN01072 PK analysis performed at cycle 1, as pre-specified according to study protocol and the data analysis plan.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 23
mcg | 141 (65.9)

19. Secondary Outcome: Fraction of IPN01072 Excreted Into the Urine (Fe) in Cycle 1
Description: as for outcome 18
Time Frame: 0 to 4 hours, 4 to 24 hours, 24 to 48 hours in Cycle 1 in Part B
Population: The IPN01072 PK set in urine (Part B only) included all participants in the ITT set who received at least 1 dose of study medication and had no major protocol deviations affecting the urine PK variables and who had all urine IPN01072 levels available to estimate the main urine PK parameters. Results were combined for IPN01072 PK analysis performed at cycle 1, as pre-specified according to study protocol and the data analysis plan.
Measure: Mean (Standard Deviation); unit: percentage of drug excreted into urine
Arm/Group | Part B: All Participants
Number analyzed (Participants) | 23
percentage of drug excreted into urine | 52.9 (24.2)

20. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR was defined as the percentage of participants who achieved a complete response (CR) or a partial response (PR) as best overall response (BOR) according centralized to response evaluation criteria in solid tumours (RECIST) version 1.1 from investigator assessment. Participants with no tumour assessment after the start of study treatment were not evaluated. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the start of the first study medication (Cycle 1 Day 1) up to 2 years after the EOCT/death or lost to follow-up, maximum of 59 months.
Population: The ITT included all participants in the eligible participants set who received study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
percentage of participants | 40.0 [16.3 to 67.7] | 16.7 [0.4 to 64.1] | 22.2 [2.8 to 60.0] | 40.0 [12.2 to 73.8] | 32.5 [18.6 to 49.1]

21. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who achieved a CR, a PR or a stable disease (SD) as BOR according to Investigator assessment RECIST version 1.1 criteria. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 20
Population: The ITT included all participants in the eligible participants set who received study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
percentage of participants | 93.3 [68.1 to 99.8] | 100.0 [54.1 to 100.0] | 100.0 [66.4 to 100.0] | 90.0 [55.5 to 99.7] | 95.0 [83.1 to 99.4]

22. Secondary Outcome: Best Overall Response
Description: The BOR according to RECIST v1.1 was defined as the best response recorded from the initiation of treatment until the EOCT/end of additional cycles (EOAC)/early withdrawal (EW) Visit (during the core study part), prior to the Investigator assessment of PD. Progression was defined as at least 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm.
Time Frame: as for outcome 20
Population: The ITT included all participants in the eligible participants set who received study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 15 | 6 | 9 | 10 | 40
Participants
  PR | 6 | 1 | 2 | 4 | 13
  SD | 8 | 5 | 7 | 5 | 25
  PD | 1 | 0 | 0 | 0 | 1
  Not Evaluable (NE) | 0 | 0 | 0 | 1 | 1

23. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as the time from start of study treatment until occurrence of tumour progression or death, according to Investigator assessment RECIST version 1.1. Estimation of the median was based on the Kaplan-Meier method.
Time Frame: as for outcome 20
Population: The ITT included all participants in the eligible participants set who received study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 6 | 3 | 6 | 5 | 20
months | 29.7 [17.5 to NA] — NA indicates upper limit of confidence interval (CI) was not evaluable due to insufficient number of participants with events. | 21.2 [19.4 to 22.4] | 25.1 [5.1 to NA] — NA indicates upper limit of CI was not evaluable due to insufficient number of participants with events. | 11.1 [5.1 to NA] — NA indicates upper limit of CI was not evaluable due to insufficient number of participants with events. | 28.1 [20.0 to NA] — NA indicates upper limit of CI was not evaluable due to insufficient number of participants with events.

24. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Questionnaire (QLQ)-C30 at EOCT Visit
Description: The European Organisation for Research and Treatment of Cancer (EORTC) score questionnaire (QLQ-C30) was used for QoL evaluation. Each scale in the questionnaire were scored (0 to 100) according to the EORTC recommendations in the EORTC QLQ-C30 scoring manual. The scale included a global health status, where high score for the global health status represents a high QoL. The functional scales consisted of physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning, where a higher value reflects a better level of function. Nine symptoms scales included nausea and vomiting, pain, fatigue, dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties, where a higher value reflects worse symptoms. Baseline was defined as the last non-missing measurement collected prior to the first dose of study drug (Day 1).
Time Frame: Baseline (Day 1) and EOCT visit (30 months)
Population: The ITT included all participants in the eligible participants set who received study medication. Only data from the participants analyzed were reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 1 | 8 | 4 | 26
score on a scale
  Global Health Status | 1.27 (23.54) | 16.70 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -6.24 (14.61) | 29.15 (28.43) | 3.84 (23.83)
  Physical functioning | -2.05 (11.03) | 0.00 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -0.82 (6.61) | 10.00 (20.00) | 0.26 (11.70)
  Role functioning | 3.85 (29.79) | 0.00 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -0.01 (19.90) | 12.50 (25.00) | 3.85 (25.08)
  Emotional functioning | 11.52 (30.15) | -25.00 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -4.16 (7.74) | 10.43 (12.51) | 5.12 (23.70)
  Cognitive functioning | 6.41 (19.89) | 0.00 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -6.26 (12.43) | 12.50 (15.95) | 3.20 (17.66)
  Social functioning: number analyzed (Participants) | 13 | 1 | 8 | 4 | 1
  Social functioning | 15.38 (33.65) | 0.00 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -2.09 (5.90) | 12.50 (25.00) | 8.97 (26.35)

25. Secondary Outcome: Change From Baseline in QLQ Gastro-intestinal. Neuroendocrine Tumour (GI.NET)21 at EOCT Visit
Description: The GI.NET21 module was intended for use among participants with gastrointestinal related (GI.- related) neuroendocrine tumours, who vary in disease stage and treatments. The module comprises 21 questions, consisting of 5 scales (endocrine symptoms, G.I. symptoms, treatment related symptom, social function, disease related worries) and 4 single items that assessed muscle /bone pain symptom, sexual function, information/communication function, and body image. Each question was quoted from 1 (not at all) to 4 (very much). Each scale in the questionnaire was scored from 0 to 100. A higher value was equivalent to worse or more problems. Baseline was defined as the last non-missing measurement collected prior to the first dose of study drug (Day 1).
Time Frame: Baseline (Day 1) and EOCT visit (30 months)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
Number analyzed (Participants) | 13 | 1 | 8 | 4 | 26
score on a scale
  Endocrine symptoms | -5.12 (13.31) | 11.10 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -0.00 (5.93) | -5.55 (11.10) | -2.98 (11.13)
  G. I. symptoms | -3.58 (13.49) | -6.70 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | 2.50 (7.04) | -13.30 (17.22) | -3.33 (12.81)
  Treatment related symptom | 5.62 (21.47) | -6.70 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | 9.01 (15.11) | -0.30 (8.15) | 5.28 (17.56)
  Social function | -19.67 (15.83) | -22.30 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | -4.15 (8.29) | -30.53 (5.55) | -16.67 (15.17)
  Disease related worries | -8.98 (14.63) | -22.20 (NA) — NA indicates that standard deviation could not be calculated as only 1 participant was analyzed. | 3.46 (16.53) | -18.05 (13.87) | -7.06 (16.37)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of the first study medication (Cycle 1 Day 1) up to 6 months after the last dose of study medication, a maximum of 33 months.
Description: The SAS included all participants who received study medication. Participants who received the therapeutic dose of 177Lu-IPN01072 during the core trial period in Part A and B.
Arm/Group | Part A: 177Lu-IPN01072 4.5 GBq | Part B Cohort 1: 177Lu-IPN01072 6 GBq | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq | All Participants
All-Cause Mortality (participants affected / at risk) | 2/15 | 0/6 | 0/9 | 1/10 | 3/40
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/6 | 2/9 | 3/10 | 8/40
Other Adverse Events (participants affected / at risk) | 15/15 | 6/6 | 9/9 | 10/10 | 39/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 177Lu-IPN01072 4.5 GBq (N=15) | Part B Cohort 1: 177Lu-IPN01072 6 GBq (N=6) | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq (N=9) | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq (N=10) | All Participants (N=40)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Precursor B-Lymphoblastic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tumour Marker Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 177Lu-IPN01072 4.5 GBq (N=15) | Part B Cohort 1: 177Lu-IPN01072 6 GBq (N=6) | Part B Cohort 3: 177Lu-IPN01072 4.5 GBq (N=9) | Part B Cohort 6: 177Lu-IPN01072 4.5 GBq (N=10) | All Participants (N=40)
Nausea (Gastrointestinal disorders) | 12 (24) | 1 (1) | 5 (13) | 8 (15) | 26 (53)
Diarrhoea (Gastrointestinal disorders) | 8 (18) | 1 (1) | 6 (14) | 6 (8) | 21 (41)
Vomiting (Gastrointestinal disorders) | 5 (8) | 0 (0) | 4 (12) | 6 (9) | 15 (29)
Abdominal Pain (Gastrointestinal disorders) | 5 (7) | 1 (1) | 1 (2) | 3 (4) | 10 (14)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (5) | 8 (11)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal Faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breath Odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent Bowel Movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia Oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Steatorrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 3 (3) | 2 (5) | 5 (11) | 13 (22)
Fatigue (General disorders) | 9 (13) | 0 (0) | 3 (6) | 1 (1) | 13 (20)
Feeling hot (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (5)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sense of oppression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (14) | 2 (2) | 3 (3) | 5 (5) | 19 (24)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 0 (0) | 1 (3) | 1 (1) | 7 (11)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 6 (7)
Dysgeusia (Nervous system disorders) | 2 (4) | 0 (0) | 2 (2) | 1 (3) | 5 (9)
Lethargy (Nervous system disorders) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 3 (8)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypogeusia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (10) | 3 (13) | 1 (4) | 1 (1) | 8 (28)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 2 (6) | 1 (1) | 1 (3) | 6 (13)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (10) | 2 (2) | 0 (0) | 5 (13)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (4) | 1 (1) | 0 (0) | 4 (7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 7 (7)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Anal fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perineal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 9 (13) | 0 (0) | 2 (5) | 1 (3) | 12 (21)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 2 (5) | 0 (0) | 3 (7)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (8) | 0 (0) | 4 (14) | 0 (0) | 7 (22)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 4 (11) | 0 (0) | 5 (13)
White blood cell count decreased (Investigations) | 2 (5) | 0 (0) | 2 (6) | 0 (0) | 4 (11)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 3 (5)
Blood urea increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 2 (5)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Albumin urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bilirubin urine present (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ambulatory abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Liver function test increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 2 (5) | 1 (2) | 7 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 2 (3) | 0 (0) | 7 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 3 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Burn oesophageal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Occupational exposure to radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Product leakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to strategic reasons, the Ipsen management team decided to early terminate the D-FR-01072-001 / OPS-C-001 study. This decision was not due to any safety or tolerability concern, or any event associated with the use of the study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT02592707/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT02592707/SAP_001.pdf